CLINICAL TRIAL: NCT02912845
Title: Post-marketing Study of KamRAB Administered as a Single Dose With Active Rabies Vaccine in Children Exposed to Rabies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Collaborators: Kedrion S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KamRAB-004
Record Dates: First submitted 2016-09-18; First posted 2016-09-23 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2019-02

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 20 IU/kg KamRAB + Active Anti-Rabies Vaccine (Experimental)
  Interventions: Drug: KamRAB - HRIG

INTERVENTIONS:
Drug: KamRAB - HRIG — wound infiltration or IM injection

SUMMARY:
The primary purpose of this study is to confirm the safety of KamRAB (Human Rabies Immunoglobulin) in children ages 0 months to <17 years, when administered as part of post-Rabies Exposure Prophylaxis (PEP).

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (male and female) ages 0 months to <17 years.
* Have been exposed or possibly exposed to rabies.
* Are indicated to receive post-exposure prophylaxis (PEP) against rabies infection.
* Have documented informed consent from the child's parent(s) or legal guardian(s) and assent from the child if appropriate.

Exclusion Criteria:

* History of previous administration of rabies vaccine or human rabies immune globulin (HRIG)
* Rabies exposure or possible rabies exposure more than seven days prior to initiation of PEP, or timing of exposure unknown

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of local and systemic adverse events occurring within 14 days of KamRAB treatment | Within 14 days from treatment
Frequency and severity of local and systemic SAEs occurring within 84 days of KamRAB treatment | Within 84 days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- ACH, Little Rock, Arkansas, United States